CLINICAL TRIAL: NCT00774189
Title: An Open Label, Balanced, Randomised, Two-Treatment, Two-Period, Two-Sequence, Single-Dose, Crossover Bioavailability Study on Clarithromycin Formulations, Comparing Clarithromycin 250 mg Tablets of Ranbaxy Laboratories With Biaxin 250 mg Tablets of Abbott Laboratories in Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study of Clarithromycin 250mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 020/CLARI-250/03
Record Dates: First submitted 2008-10-15; First posted 2008-10-17 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence clarithromycin 250mg tablets fasting
MeSH Terms: interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): clarithromycin 250 mg tablets of Ranbaxy Laboratories
  Interventions: Drug: clarithromycin 250 mg tablets
- 2 (Active Comparator): Biaxin 250 mg tablets
  Interventions: Drug: clarithromycin 250 mg tablets

INTERVENTIONS:
Drug: clarithromycin 250 mg tablets

SUMMARY:
The objective of the study was to compare the single-dose oral bioavailability of Clarithromycin 250 mg tablets of Ranbaxy Laboratories with Biaxin 250 mg tablets of Abbott Laboratories in healthy, adult, human subjects under fasting conditions

DETAILED DESCRIPTION:
This was an open label, balanced, and randomized, two-treatment, two-period, two-sequence, single-dose, crossover bioavailability study planned on 32 healthy, adult, human subjects under fasting conditions. 31 subjects completed both the periods of the study. Both periods were separated by a washout of twelve days The study was conducted on 32 healthy, adult, human subjects under fasting conditions. 31 subjects completed both the periods of the study

ELIGIBILITY:
Inclusion Criteria:

1. Be in the age range of 18-45 years.
2. Be neither overweight nor underweight for his/her height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
3. Have voluntarily given written informed consent to participate in this study.
4. Be of normal health as determined by medical history and physical
5. Examination of the subjects performed .within 14 days prior to the commencement of the study.
6. If female and:

Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence; or~ Is postmenopausal for at least 1 year; or Is surgically sterile bilateral tubal ligation, bilateral oophorectomy, or hysterectomy)

Exclusion Criteria:

1. History of allergy to clarithromycin, erythromycin and related macrolides
2. Any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
3. Presence of disease markers of HIV 1 and 2, Hepatitis B and C viruses and syphilis infection.
4. Female volunteers demonstrating a positive pregnancy screen.
5. Female volunteers who are currently breastfeeding.
6. Presence of values' which are clinically significantly different from normal reference ranges for haemoglobin, total white blood cells count, differential WBC count and platelet count
7. Positive for urinary screen testing of drugs of abuse (opiates and cannabinoids
8. Presence of values which are significantly different from normal.reference ranges (as defined in Appendix 5) for se- rum creatinine, blood urea nitrogen serum aspartate aminotransferase (AST), serum alanine aminotranferase (ALT), serum alkaline phosphatase, serum billrubin, plasma glucose and serum cholesterol
9. Clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells (>4/HPF), glucose, (positive) and protein (positive).
10. History of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or hematological disease, diabetes or glaucoma.
11. History of any psychiatric illness. which may impair the ability to provide written informed consent.
12. Regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
13. History of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 'unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
14. Use of any enzyme modifying drugs within 30 days prior to Day I of this study
15. Participation in any clinical trial within 12 weeks preceeding day 1 of study
16. Subjects who, through completion of this study, would have donated and/or lost more than 350 mL of blood in past 3 months

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-07; Primary Completion 2003-08 (Actual); Study Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Ranbaxy Research Laboratories, Gurgaon, Haryana, India

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm